CLINICAL TRIAL: NCT03309085
Title: Functional Imaging With Computational Fluid Dynamics to Evaluate the Airways in Patients With Acute Lung Injury
Brief Title: Functional Respiratory Imaging of Airways in ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Tom Schepens, MD, Research fellow, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: EC 10/52/359; B300201010195 (Registry Identifier: Belgian national registry)
Record Dates: First submitted 2017-10-03; First posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Repeated CT scan
  Interventions: Procedure: Repeated CT scan; Device: CT scan

INTERVENTIONS:
Procedure: Repeated CT scan — CT scan of chest on different PEEP levels, 4 in total
Device: CT scan — CT scan

SUMMARY:
This is a prospective single-center cohort trial to compare regional bronchial recruitment, bronchial distention and alveolar recruitment in 6 patients with acute respiratory distress syndrome (ARDS). The investigators used CT scan images as the imaging modality, and the subjects were scanned on end-expiratory lung volume with different positive end-expiratory pressures. Those images were post-processed to evaluate the airways.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated
* moderate or severe ARDS, as defined by the Berlin criteria

Exclusion Criteria:

* pregnancy
* hemodynamic instability
* obesity (BMI >30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2014-04-14 (Actual); Study Completion 2014-04-14 (Actual)

PRIMARY OUTCOMES:
Regional bronchial recruitment | Through study completion, within 24 hours after inclusion
  The difference in bronchial tree volume increase from one PEEP level to the other
Regional bronchial dilation | Through study completion, within 24 hours after inclusion
  The difference in bronchial diameter from one PEEP level to the other
Regional alveolar recruitment | Through study completion, within 24 hours after inclusion
  The difference in alveolar volume from one PEEP level to the other

SECONDARY OUTCOMES:
Correlation between parenchymal recruitment and bronchial recruitment | Through study completion, within 24 hours after inclusion
  Correlation between parenchymal recruitment (in milliliter) and bronchial (in milliliter) recruitment for each type of ARDS (focal versus diffuse)

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No